CLINICAL TRIAL: NCT00800943
Title: A Clinical Research Consortium (CRC) Phase II Study of Subcutaneous Campath-1H in Patients With B-Cell Chronic Lymphocytic Leukemia and Residual Disease After Chemotherapy
Brief Title: Study of Subcutaneous Campath-1H in Patients With B-Cell CLL and Residual Disease After Chemotherapy
Acronym: CRC005
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chronic Lymphocytic Leukemia Research Consortium (Network)
Collaborators: Bayer (Industry)
Responsible Party: Thomas J. Kipps, M.D., Ph.D., University of California, San Diego, CLL Research Consortium
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRC005
Record Dates: First submitted 2008-12-01; First posted 2008-12-03 (Estimated); Last update posted 2008-12-03 (Estimated); Status verified 2008-12

CONDITIONS: B-Cell Chronic Lymphocytic Leukemia
Keywords: Leukemia; Chronic; Chronic Lymphocytic Leukemia; CAMPATH; Alemtuzumab; MabCampath; Subcutaneous; CLL; C-CLL; Residual
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia; Bronchiolitis Obliterans Syndrome | interventions — Alemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Campath-1H (Experimental)
  Interventions: Biological: Alemtuzumab (Campath-1H)

INTERVENTIONS:
Biological: Alemtuzumab (Campath-1H) — Campath is administered using escalating doses and alternating injection sites. The dose is escalated as tolerated using 3mg,10mg,and 30mg, administered subcutaneously (SC) (if tolerated). When escalation to 30 mg dose is tolerated, all subsequent doses are administered at 30 mg SC 3 times per week at alternating injection sites for up to 8 weeks

SUMMARY:
To evaluate whether CAMPATH-1H given to patients with CLL after maximum response to chemotherapy will: a) eliminate minimal residual disease (documented by flow cytometry) in patients who have achieved a complete remission (CR) or b) convert partial remission to complete remission.

To evaluate the time-to-progression of patients according to pretreatment characteristics and response status at study entry.

To evaluate whether CAMPATH-1H given to patients with CLL after maximum response to chemotherapy will eliminate minimal residual disease as determined by real-time quantitative PCR.

DETAILED DESCRIPTION:
Approximately 95% of cases involve the clonal proliferation of B cells. Paraproteins, often of the IgM class, can be detected in the serum and/or urine of most patients with CLL. Unique cell surface markers are increasingly being used to diagnose the disease, and in approximately 40% of patients, cytogenetic abnormalities (for example, trisomy 12) can be found. Patients commonly present with lymphocytosis, lymphadenopathy, splenomegaly and symptoms of fatigue, weight loss, and malaise. In more advanced cases anemia and thrombocytopenia can also occur. The clinical course of CLL is unpredictable, with survival from initial diagnosis varying from 1 to 20 years (2). In addition, there is a subset of patients with indolent CLL whose absolute lymphocyte count is less than 30 x 109/L and who rarely die from the disease.

CLL is commonly staged according to the 5-point system proposed by Rai (Appendix B) and co-workers. While Rai staging is a relatively good predictor of overall survival, it cannot predict the prognosis in individual patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, at least 18 years old.
* Signed informed consent.
* Zubrod performance status of 0, 1, or 2 (Appendix C).
* Patients with CLL, CLL/PLL or PLL (prolymphocytic) who have achieved a clinical complete remission by NCI-WG criteria with chemotherapy, eg., alkylating agents, fludarabine or chemoimmunotherapy but have documentation of residual disease by immunophenotyping showing: (a) a residual population of CD5 and CD19 positive cells that comprise ≥ 10% of the marrow mononuclear cell population; or (b) a residual population of CD5 and CD19 positive cells that comprise <10% of the marrow mononuclear cells and have a Kappa/Lambda ratio >6 or <.33.
* Patients with CLL who have achieved a partial remission (PR) or nodular partial remission (nPR) by NCI-WG criteria after chemotherapy.
* Creatinine, bilirubin, AST or ALT and alkaline phosphatase ≤2 x the upper limit of normal.

Exclusion Criteria:

* Active infection.
* Past history of anaphylaxis, following exposure to rat or mouse derived CDR-grafted humanized monoclonal antibodies.
* Less than 2 months since prior chemotherapy.
* Previous treatment with CAMPATH-1H.
* Pregnant or nursing women.
* Patients on corticosteroids.
* Uncontrolled autoimmune hemolytic anemia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2003-12; Primary Completion 2010-08 (Estimated); Study Completion 2010-08 (Estimated)

PRIMARY OUTCOMES:
To evaluate whether CAMPATH-1H given to patients with CLL after maximum response to chemotherapy will: a) eliminate residual disease (documented by flow cytometry) or b) convert partial remission to complete remission | Response evaluation at end of each course (4 weeks of therapy) (within 0-8 weeks). Patients followed until progressive disease is documented or death

SECONDARY OUTCOMES:
To evaluate the time-to-progression of patients according to pretreatment characteristics and response status at study entry. | Response evaluation at end of each course (4 weeks of therapy) (within 0-8 weeks). Patients followed until progressive disease is documented or death.
To evaluate whether CAMPATH-1H given to patients with CLL after maximum response to chemotherapy will eliminate minimal residual disease as determined by real-time quantitative PCR. | Response evaluation at end of each course (4 weeks of therapy) (within 0-8 weeks). Patients followed until progressive disease is documented or death.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Kipps, MD, PhD, Principal Investigator — Director, Chronic Lymphocytic Leukemia Research Consortium
Locations (3):
- United States (3):
  - University of California San Diego, La Jolla, California
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - M. D. Anderson Cancer Center at University of Texas, Houston, Texas